CLINICAL TRIAL: NCT02257151
Title: Randomized, Double-Blind, Placebo-Controlled, Single and Multiple Ascending Dose Study to Evaluate the Safety, and Pharmacokinetics of BMS-986142 in Healthy Subjects
Brief Title: Study to Evaluate the Safety, Pharmacokinetics and Target Engagement of BMS-986142 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IM006-001
Record Dates: First submitted 2014-10-02; First posted 2014-10-06 (Estimated); Last update posted 2015-09-24 (Estimated); Status verified 2015-09

CONDITIONS: Healthy Adult
Keywords: Volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1: BMS-986142 or placebo (Experimental): BMS-986142 or placebo Single dose oral Solution or spray dried dispersion as specified
  Interventions: Drug: BMS-986142; Drug: Placebo
- Group 2: BMS-986142 or placebo (Experimental): BMS-986142 or placebo Multiple dose oral Solution as specified
  Interventions: Drug: BMS-986142; Drug: Placebo

INTERVENTIONS:
Drug: BMS-986142
Drug: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, pharmacokinetics, and target engagement of BMS-986142 in healthy subjects.

DETAILED DESCRIPTION:
Allocation: Randomized Controlled Trial (SAD/MAD) Masking: Double-Blind (SAD/MAD)

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

1. Healthy male and female subjects as determined by no clinically significant deviation from normal in medical history, physical examination, ECGs, and clinical laboratory determinations
2. Body Mass Index (BMI) of 18 to 32 kg/m2, inclusive. BMI=weight (kg)/[height(m)]2

Exclusion Criteria:

1. Any significant acute or chronic medical illness
2. Current or recent (within 3 months of study drug administration) gastrointestinal disease
3. Any major surgery within 4 weeks of study drug administration
4. Any gastrointestinal surgery that could impact upon the absorption of study drug
5. Donation of blood to a blood bank or in a clinical study (except a screening visit) within 4 weeks of study drug administration (within 2 weeks for plasma only)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 118 (Actual)
Dates: Start 2014-09; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Primary safety endpoint is based on the incidence, potential significance, and clinical importance of adverse events after single dose of BMS-986142 | Single Ascending Dose(SAD) within 8 days
Primary safety endpoint is based on the incidence, potential significance, and clinical importance of adverse events after multiple doses of BMS-986142 | Multiple Ascending Dose (MAD) within 19 days

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Wcct Global, Llc, Cypress, California, United States

REFERENCES:
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx